CLINICAL TRIAL: NCT02103673
Title: DAOIB for the Treatment of Cognitive Function and Behavioral and Psychological Symptoms of Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chieh-Hsin Lin, Dr, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 102-0035C
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Behavioral and Psychological Symptoms in Alzheimer's Disease; Behavioral and Psychological Symptoms in Vascular Dementia
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- DAOIB (Experimental): Drug: DAOIB 250-1500 mg/day by mouth for 6 weeks
  Interventions: Drug: DAOIB
- Placebo (Placebo Comparator): Placebo by mouth per day for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DAOIB — Intervention drug: DAOIB. Dosage: 250-1500 mg/day by mouth. Duration: 6 weeks
  Arms: DAOIB
Drug: Placebo — Intervention drug: placebo by mouth. Duration: 6 weeks
  Arms: Placebo

SUMMARY:
The population of dementia is increasing rapidly. Cognitive impairment as well as Behavioral and psychological symptoms of dementia (BPSD) add heavy burdens to caregiver. NMDA activation is critical for learning and memory. Individuals with Alzheimer's disease (AD) have fewer NMDA receptors in the frontal cortex and hippocampus than controls. This study is a randomized, double-blind, placebo-controlled drug trial. All patients will be allocated randomly to two groups: (1) NMDA enhancer: DAOIB (starting dosage: 250-500 mg/day), (2) placebo, for 6 weeks. The investigators hypothesize that DAOIB may yield better efficacy than placebo for cognitive function and clinical symptoms in patients with BPSD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of probable Alzheimer's disease or probable vascular dementia
* For patients with vascular dementia, the post-stroke period must be more than 3 months
* Mini-Mental State scores between 5-26
* Clinical Dementia Rating score equal to or greater than 1
* Behavioral Pathology in Alzheimer's Disease Rating Scale score equal to or greater than 2

Exclusion Criteria:

* Current substance abuse or history of substance dependence in the past 6 months
* Other major psychiatric diagnoses, such as schizophrenia, major depressive disorder, bipolar disorder and mental retardation etc.
* Serious medical or neurological illness other than Alzheimer's disease/vascular dementia and other secondary dementia

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-02; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Behavioral Pathology in Alzheimer's Disease Rating Scale | weeks 0, 2, 4, 6
  Change from baseline in Behavioral Pathology in Alzheimer's Disease Rating Scale at weeks 2, 4 and 6
Alzheimer's Disease Assessment Scale - cognitive subscale | weeks 0 and 6
  Change from baseline in Alzheimer's Disease Assessment Scale - cognitive subscale at week 6

SECONDARY OUTCOMES:
Neuropsychiatirc Inventory | weeks 0 and 6
  Change from baseline in Neuropsychiatirc Inventory at week 6
Instrumental Activities of Daily Living | weeks 0 and 6
  Changes from baseline in Instrumental Activities of Daily Living at week 6
Zarit Caregiver Burden Interview | weeks 0 and 6
  Changes from baseline in Zarit Caregiver Burden Interview at week 6
Geriatric Geriatric Depression Scale | weeks 0, 2, 4, 6
  Changes from baseline in Geriatric Depression Scale at weeks 2, 4 and 6
Mini-Mental Status Examination | weeks 0 and 6
  Changes from baseline in Mini-Mental Status Examination at week 6

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-Yuan Lane, MD, PhD, Study Chair — China Medical University Hospital
Locations (2):
- Taiwan (2):
  - Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung

REFERENCES:
- [Derived] Lin CH, Chen PK, Wang SH, Lane HY. Effect of Sodium Benzoate on Cognitive Function Among Patients With Behavioral and Psychological Symptoms of Dementia: Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2021 Apr 1;4(4):e216156. doi: 10.1001/jamanetworkopen.2021.6156. PMID 33881530
- [Derived] Lin CH, Yang HT, Chen PK, Wang SH, Lane HY. Precision Medicine of Sodium Benzoate for the Treatment of Behavioral and Psychological Symptoms of Dementia (BPSD). Neuropsychiatr Dis Treat. 2020 Feb 20;16:509-518. doi: 10.2147/NDT.S234371. eCollection 2020. PMID 32110025